CLINICAL TRIAL: NCT05091645
Title: Translation and Cultural Adaptation of the Greek Version of the Groningen Frailty Indicator (GFI) in Patients With Hip Fracture; a Prospective Cohort Study
Brief Title: Translation and Cultural Adaptation of the Groningen Frailty Indicator (GFI) in Patients With Hip Fracture
Acronym: Gr-GFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: Gr-Groningen Frailty Indicator
Record Dates: First submitted 2021-10-21; First posted 2021-10-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Frailty Syndrome; Hip Fractures
Keywords: Frailty Syndrome; Hip fractures; Cultural adaptation; Translation
MeSH Terms: conditions — Frailty; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip fracture_GFI: Greek patients with hip fracture assessed for frailty syndrome with the adapted for the greek population GFI questionnaire
  Interventions: Other: GFI

INTERVENTIONS:
Other: GFI — Two trained raters who will be blinded and will have no access to each other's evaluation, will administer the GFI questionnaire within 24 hours of patients' hospital admission.

SUMMARY:
This study attempts to the translation and the cultural adaptation of the Groningen Frailty Indicator (GFI) questionnaire in the Greek population in patients suffering from hip fracture.

DETAILED DESCRIPTION:
Frailty indicates a state of vulnerability in terms of poor health outcomes, such as mortality, hospitalization, institutionalization and loss of function in one or more domains (i.e. physical, psychological, cognitive and social domains). Frailty is not only associated with poor quality of life and life satisfaction but also has an effect on health care demands, as the number of frail people in our aging population will increase.

Current literature suggests that frailty is a common condition among elderly patients with hip fracture. Ageing has been associated with a decline in physiological reserves which impedes the body's ability to withstand and recover from minor and major challenges, such as the hip fracture. Hence, accurate diagnosis of frailty seems mandatory. The Groningen Frailty Indicator (GFI) questionnaire is a feasible, reliable and valid self-assessment tool.

This study will provide the first official Greek translation and cultural adaptation of the GFI according to the ISPOR (International Society for Pharmacoeconomics and Outcomes Research) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over 65 years old with hip fractures undergoing surgery
* an ASA (American Society of Anesthesiologists) PS (physical status) I to III
* non-institutionalized
* able to communicate orally or in writing
* consent to participate

Exclusion Criteria:

* refused to participate
* pathological hip fractures
* institutionalized
* patients with hip fracture treated conservatively
* patients with severe cognitive dysfunction
* patients with insufficient knowledge of the Greek language

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with hip fractures undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Translation and Cultural adaptation of the Greek version of Groningen Frailty Indicator (GFI) questionnaire | Within 24 hours of the hospital admission
  Translation and Cultural adaptation of the Greek version of GFI

SECONDARY OUTCOMES:
Incidence of frailty syndrome | Baseline (On admission)
  Incidence of frailty syndrome in our study sample

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Principal Investigator — University of Thessaly; Michael Hantes, MD, PhD, Principal Investigator — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No